CLINICAL TRIAL: NCT03500796
Title: Combined Amniotic Membrane and Platelet Rich Plasma Clot for Management of Central Corneal Perforation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahemd Abdelghany, Lecturer of Ophthalmology, Faculty of Medicine, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 56-2/2018
Record Dates: First submitted 2018-03-23; First posted 2018-04-18 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Corneal Perforation
MeSH Terms: conditions — Corneal Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corneal perforation patients (Other): Patients who had/impeding corneal perforation due to melting of the cornea after infection with a corneal pathogen (bacterial or viral), with no previous surgical intervention.
  Patients will undergo:
  Platelet rich plasma clot implantation Wound closure with amniotic membrane
  Interventions: Procedure: Platelet rich plasma clot implantation; Procedure: Wound closure with amniotic membrane

INTERVENTIONS:
Procedure: Platelet rich plasma clot implantation — Implantation of a platelet rich plasma clot, which is created from the plasma of the patients, and refrigerated to be inserted under the sealing amniotic membrane
Procedure: Wound closure with amniotic membrane — Closure of the corneal perforation with a synthetic amniotic membrane with a 2 mm safety margin

SUMMARY:
Use of amniotic membrane(AMT) and platelet rich plasma (PRP) clot for closure of central corneal perforation

DETAILED DESCRIPTION:
Use of amniotic membrane and platelet rich plasma clot for closure of central corneal perforation either post infective or posttraumatic

ELIGIBILITY:
Inclusion Criteria:

* central corneal perforation

Exclusion Criteria:

* active infection
* posterior segment pathology
* non seeing eye

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Closure of the corneal wound | 3 months
  sealing of the edges corneal gap, with formation of scar tissue

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Abdelghany, MD, Principal Investigator — Assistant professor of Ophthalmology, Faculty of Medicine
Locations (1):
- Faculty of Medicine, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No
steps of technique and results